CLINICAL TRIAL: NCT00002245
Title: Effect of Amprenavir on Carbohydrate and Lipid Metabolism in Patients With HIV Infection
Brief Title: A Study of the Effects of Amprenavir, a Protease Inhibitor, on Carbohydrate and Fat Metabolism in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 264L; COL30309
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Lamivudine; Carbohydrates; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Lipids; Insulin Resistance; abacavir
MeSH Terms: conditions — HIV Infections; Insulin Resistance | interventions — abacavir; amprenavir; Lamivudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Lamivudine

SUMMARY:
The purpose of this study is to evaluate the effects of a 3-drug anti-HIV regimen, amprenavir (APV) plus abacavir (ABC) plus lamivudine (3TC), on the way carbohydrates (sugars) and fats are metabolized (processed by the body) in HIV-infected patients who have received little or no previous anti-HIV drug therapy.

DETAILED DESCRIPTION:
This single-site study uses an open-label, single-arm design to evaluate the effects of APV, a protease inhibitor (PI), plus concurrent nucleoside reverse transcriptase inhibitors (NRTIs) ABC and 3TC on carbohydrate and lipid metabolism in non-diabetic, HIV-1 infected patients initiating antiretroviral therapy. Treatment duration is 24 weeks, and patients serve as their own controls. The combination therapy is evaluated for safety, tolerability, efficacy, and effects on body composition. The proportion of patients who attain plasma HIV RNA below the lower limit of quantitation of the Roche Amplicor (less than 400 copies/ml) and Ultrasensitive (less than 50 copies/ml) is measured at 24 weeks after starting therapy with APV plus ABC plus 3TC.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years old.
* Have very little or no anti-HIV drug experience (see below for details) and have never taken ABC.
* Have a CD4 count greater than or equal to 200 cells/mm3 within 30 days prior to study entry.
* Have a viral load (level of HIV in the blood) greater than 500 copies/ml within 30 days prior to study entry.
* Agree to use effective methods of birth control during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken both 3TC and stavudine (d4T).
* Have taken a protease inhibitor (PI) or nonnucleoside reverse transcriptase inhibitor (NNRTI) for more than 7 days.
* Have taken a PI within 60 days of study entry.
* Have a history of diabetes.
* Have a history of untreated gonad or thyroid disorder.
* Have a stomach or intestinal disorder which may affect the way the body absorbs the study drugs, or which may make them unable to take medications by mouth.
* Have received chemotherapy or radiation within 4 weeks prior to entry, or if they will need either of these during the study period.
* Have lost or gained a significant amount of weight (greater than 5%) within the past 2 months.
* Have a serious medical condition, such as heart disease.
* Are allergic to any of the study drugs.
* Have been treated for an infection or other medical illness within 14 days prior to study entry.
* Have had a fever (over 38.5 degrees Celsius) for any 7 days or chronic diarrhea (more than 3 liquid stools per day for 15 days) within 30 days prior to study entry.
* Have an AIDS-related cancer (other than Kaposi's sarcoma).
* Abuse alcohol or drugs.
* Have received certain medications.
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: M Dube, Study Chair
Locations (1):
- LAC / USC Med Ctr / Infectious Diseases, Los Angeles, California, United States